CLINICAL TRIAL: NCT07085364
Title: Attentional Focus Training on Visuomotor Control in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20250107004
Record Dates: First submitted 2025-06-05; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Gait; Attention; Older Adults
Keywords: attentional focus; gait; visual search; older adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXT (Experimental): External focus manipulation
  Interventions: Behavioral: Attentional focus
- CON (Active Comparator): Traditional manipulation
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Attentional focus — Every training session will include the following activities for both groups: a 5-minute warm-up; a 30-minute walking training; and a 5-minute cool-down. The walking training will be conducted within a level-ground walking field. Participants will be instructed to look at and step on specific markers/labels that will be attached along the walking paths.
  Arms: EXT
Behavioral: Control — Every training session will include the following activities for both groups: a 5-minute warm-up; a 30-minute walking training; and a 5-minute cool-down. The walking training will be conducted within a level-ground walking field. No markers/labels will be attached and no relevant instructions will be provided apart from the general instruction.
  Arms: CON

SUMMARY:
This study will be a pilot randomized controlled trial, to investigate the effectiveness of an external focus training on visuomotor performance while comparing with an active control group.

DETAILED DESCRIPTION:
All eligible participants will be randomly divided into two groups: external focus gait training group (EXT) and active control group (CON). All participants will complete two assessment sessions: at baseline (T0) and immediately following the completion of all training sessions (T1). A total of twelve training sessions (about 45 minutes per session), held twice a week for six weeks, would be provided to participants in both training groups.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 or above
* able to walk independently indoor for at least 40 metres
* static visual acuity score 20/40 or above
* scoring 22/30 or above in the Montreal Cognitive Assessment Hong Kong version
* without any history of untreated major neurological, vestibular or musculoskeletal deficits (e.g., stroke or Parkinson's disease)
* without any unstable medical condition that can compromise safety during the experiment
* scoring less than 24/28 in the Tinetti Balance Assessment Tool or scoring 50/56 or below in the Berg Balance Scale

Exclusion Criteria:

* none

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Gait stability - variability of stride time | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by a 3-D motion capture system; stride time is defined as the interval between two consecutive heel strikes of the same foot; the variability measure is represented by the coefficients of variation (CV) [(standard deviation/mean) × 100]
Gait stability - variability of stride length | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by a 3-D motion capture system; stride length is defined as anterior-posterior (A-P) distance between two consecutive heel strike positions of the same foot; the variability measure is represented by the coefficients of variation (CV) [(standard deviation/mean) × 100]
Gait stability - variability of step width | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by a 3-D motion capture system; step width is defined as medial-lateral (M-L) distance between two consecutive heel strike positions of the opposite feet; the variability measure is represented by the coefficients of variation (CV) [(standard deviation/mean) × 100]
Visual search behaviours - location of fixation | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by a wireless eye tracker; recorded the location that the gaze is fixated on
Visual search behaviours - the number of fixation | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by a wireless eye tracker; recorded the number of times the gaze is fixated on each area of interest
Visual search behaviours - fixation duration | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by a wireless eye tracker; recorded the duration that the gaze is fixated on each area of interest

SECONDARY OUTCOMES:
Functional balance and gait | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by the Tinetti Balance Assessment Tool; min: 0; max: 28; higher scores reflect better functional balance and gait
Falls efficacy | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by the Chinese version of the Falls Efficacy Scale International; min: 16; max: 64; higher scores reflect greater concern about falling
Conscious movement processing | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by the Chinese version of the Movement Specific Reinvestment Scale; min: 10, max: 60; higher scores reflect higher propensity for conscious movement processing
Functional balance | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by the Berg Balance Scale; min: 0; max: 56; higher scores reflect better functional balance
Functional mobility | baseline (pre-intervention), immediately after intervention (post-intervention)
  measured by the Timed 'Up & Go' Test (in seconds); a longer time to complete reflects poorer functional mobility

IPD SHARING:
Plan to Share IPD: No